CLINICAL TRIAL: NCT01173302
Title: Persistence of Rabies Antibody 1-5 Years After the Post-exposure Prophylaxis With Vero Cell Antirabies Vaccine and Antibody Response to a Single Booster Dose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Dr. Wang Chuanlin, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PKUPH-ER-1
Record Dates: First submitted 2010-07-19; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Rabies
Keywords: Rabies; Anti-rabies antibody; Persistence
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Post vaccination (Experimental): All the subjects had been vaccinated with antirabies vaccine.
  Interventions: Biological: Rabies vaccine, manufactured by ChengDa

INTERVENTIONS:
Biological: Rabies vaccine, manufactured by ChengDa — 1 dose before the antibody is tested
  Other Names: ChengDa Speeda

SUMMARY:
This study is to investigate the persistence of rabies Chinese manufactured antibody 1-5 years after the post-exposure prophylaxis with vero cell antirabies vaccine and antibody response to a single booster dose. A total of 160 subjects would be enrolled. These subjects were all administered ChengDa antirabies vaccine from 2005 to 2009. After informed consent is obtained, these subjects would be tested for their antirabies antibody titer and given a single booster dose. Seven and 14 days later, the investigators would re-evaluate the antibody titer.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 60 years old
* Healthy
* Given ChengDa rabies vaccine
* Good compliance
* Obtained informed consent

Exclusion Criteria:

* Other than inclusion criteria

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Rabies antibody titer | 6 months
  We test the antirabies antibody titer before and after the single booster dose

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang X, Zhu Z, Wang C. Persistence of rabies antibody 5 years after postexposure prophylaxis with vero cell antirabies vaccine and antibody response to a single booster dose. Clin Vaccine Immunol. 2011 Sep;18(9):1477-9. doi: 10.1128/CVI.05090-11. Epub 2011 Jul 13. PMID 21752947